CLINICAL TRIAL: NCT02754700
Title: Effects of Real-time Optimized Biofeedback Utilizing Sport Techniques (ROBUST) Training on Risk of Anterior Cruciate Ligament Injury
Brief Title: Real-time Optimized Biofeedback Utilizing Sport Techniques
Acronym: ROBUST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: High Point University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AR069873 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Knee Injuries
Keywords: Anterior Cruciate Ligament
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biofeedback Hip (Experimental): Hip focused biofeedback with neuromuscular training
  Interventions: Other: Hip Focused ROBUST Training
- Biofeedback Knee (Experimental): Knee focused biofeedback with neuromuscular training
  Interventions: Other: Knee Focused ROBUST Training
- Neuromuscular Training (Active Comparator): Neuromuscular Training component
  Interventions: Other: Neuromuscular Training

INTERVENTIONS:
Other: Neuromuscular Training — Standardized, comprehensive neuromuscular training
  Arms: Neuromuscular Training
Other: Hip Focused ROBUST Training — Biofeedback training focused on the hip extensors
  Arms: Biofeedback Hip
Other: Knee Focused ROBUST Training — Biofeedback training focused on knee abduction
  Arms: Biofeedback Knee

SUMMARY:
This study will identify the most optimal, focused approach for biofeedback in adolescent females at high risk for anterior cruciate ligament (ACL) injury. A six-week randomized, pre/post-testing design will be used to identify biofeedback training effects. The investigators will also determine the effects of hip strategy on retention of decreased knee abduction load with focused biofeedback. A six-month follow-up design will be used to test retention of real-time biofeedback intervention.

DETAILED DESCRIPTION:
Real-time Optimized Biofeedback Utilizing Sport Techniques (ROBUST) represents an innovative new approach to reduce traumatic anterior cruciate ligament (ACL) injuries. Over the last four decades, these debilitating injuries have occurred at a 2 to 10-fold greater rate in female compared to male athletes with the highest prevalence occurring between the ages of 16-18 years. As a consequence, there is a large population of females that endure significant pain, functional limitations and knee osteoarthritis (OA) as early as 5 years after the initial unintentional injury. To reduce the burden of OA, The National Public Health Agenda for Osteoarthritis recommends both expanding and refining evidence-based prevention of ACL injury. There currently is a gap in knowledge regarding how to maximize the effectiveness of injury prevention training in young female athletes. The long-term goal is to reduce ACL injuries in young female athletes. The objective of this application is to increase the efficacy of biofeedback training to reduce the risk of ACL injury. This proposal tests the central hypothesis that biofeedback methodology is needed to maximize the effectiveness of neuromuscular prophylactic interventions. The rationale supporting this proposal is that once the proposed research is completed, health professionals will be more successful at preventing devastating ACL injuries through properly optimized and targeted biofeedback training for young at-risk females. This research is innovative because it represents a new and substantive departure from the status quo by recognizing the need to optimize the application of biofeedback training. The work will contribute clinically relevant data in support of a future more robust clinical trial. The proposed research will be significant because it will lead to reduced rates of ACL injury in young females. Reduction of female injury rates to equal that of males would allow females annually to continue the health benefits of sports participation and avoid the long-term complications of osteoarthritis, which occurs with a 10 to 100-fold greater incidence in ACL-injured than in uninjured athletes.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating on club or school sponsored soccer team

Exclusion Criteria:

* Current injury that limits participating in sport
* Male
* Cannot participate in a 6-week intervention due to time or other constraints

Ages: 9 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Knee abduction load | 6 weeks
  Knee abduction load will be the primary outcome measure. This is assessed with three-dimensional motion analysis techniques and a detailed full-body biomechanical model during dynamic landing tasks immediately before and after 6 weeks of the study intervention. The unit of measure for knee abduction load is Nm and will be normalized to participant mass when appropriate.

SECONDARY OUTCOMES:
Knee abduction load | 6 months
  Knee abduction load following a 6 month retention time will be the secondary outcome measure. This is assessed with three-dimensional motion analysis techniques and a detailed full-body biomechanical model during dynamic landing tasks following 6 months after study intervention. The unit of measure for knee abduction load is Nm and will be normalized to participant mass when appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ford, PhD, Principal Investigator — High Point University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ford KR, Taylor JB, Westbrook AE, Paterno MV, Huang B, Nguyen AD. Outcomes of a randomized controlled trial of neuromuscular training with real-time biofeedback in young female athletes. BMC Musculoskelet Disord. 2025 Apr 15;26(1):366. doi: 10.1186/s12891-025-08647-3. PMID 40234828
- [Derived] Taylor JB, Nguyen AD, Paterno MV, Huang B, Ford KR. Real-time optimized biofeedback utilizing sport techniques (ROBUST): a study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Feb 7;18(1):71. doi: 10.1186/s12891-017-1436-1. PMID 28173788